CLINICAL TRIAL: NCT01056991
Title: A Study to Determine if Modern Under-patient Warming Mattresses Are as Effective as Forced-air Warming Blankets in Preventing Peri-operative Hypothermia
Brief Title: Prevention of IPH: Electric Warming Mattress vs Forced Air Warming Blanket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr C. Mark Harper, Consultant Anaesthetist, Brighton and Sussex University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09/183/HAR
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Inadvertent Perioperative Hypothermia; Patient Warming

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- warming mattress (Experimental): Patient warmed with electric mattress
  Interventions: Other: warming mattress
- warming blanket (Active Comparator): Forced air warming blanket
  Interventions: Other: warming blanket

INTERVENTIONS:
Other: warming mattress — comparison of under patient warming mattress to forced air warming blankets in preventing peri-operative hypothermia
  Other Names: Inditherm electric carbon polymer warming mattress
  Arms: warming mattress
Other: warming blanket
  Other Names: forced-air warming blanket; Bair hugger
  Arms: warming blanket

SUMMARY:
This study will determine if modern under-patient warming mattresses are as effective as forced air warming blankets in preventing cold and shivering in patients scheduled for non emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective (non emergency) surgery who will require intra-operative warming
* Patients whose surgery will be performed with them in the supine position

Exclusion Criteria:

* Abdominal aortic aneurysm repair
* All adults (over 18 years) who refuse,who are unable to fully understand the trial
* ALL laparoscopic surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Post-operative core temperature greater than or equal to 36 degrees centigrade. This is a surrogate marker for complications such as reduced wound infection and reduced hospital stay that have been previously established by other research. | 15minutes to 2 hours approximately postoperatively in recovery room

SECONDARY OUTCOMES:
shivering | up to 2h post op (time in recovery)
Core temperature | From induction of anaesthesia to arrival in recovery

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Harper, MBBS FRCA, Principal Investigator — BSUH
Locations (1):
- Royal Sussex County Hospital, BSUH NHS Trust, Brighton, United Kingdom

REFERENCES:
- [Derived] John M, Crook D, Dasari K, Eljelani F, El-Haboby A, Harper CM. Comparison of resistive heating and forced-air warming to prevent inadvertent perioperative hypothermia. Br J Anaesth. 2016 Feb;116(2):249-54. doi: 10.1093/bja/aev412. PMID 26787794